CLINICAL TRIAL: NCT06633549
Title: Investigation of the Effect of Home Accidents Prevention Training Given to Mothers of Mentally Disabled Children Aged 0-6: A Randomized Controlled Trial
Brief Title: The Effect of Home Accidents Prevention Training Given to Mothers of Mentally Disabled Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Principal Investigator, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022/21-07
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Mental Disability; Mothers; Home Injury
Keywords: home accidents; child; mother; risk factors; mental disability
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educated (Experimental): Educated Group
  Interventions: Other: Home Accidents Prevention Training
- Uneducated (Other): Uneducated Group (Control)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Home Accidents Prevention Training — Mothers in the education group who participated in the study were informed about the research and their written consent was obtained. Mothers filled out the 'Information Form' then completed the 'Diagnostic Scale of the Mother's Safety Measures for Home Accidents in Children Aged 0-6 Years'. Mothers were helped when filling out the form and their questions were answered. The training program was organized so that there would be a maximum of 5 mothers in each group. The trainings were conducted face-to-face with a PowerPoint presentation and lasted about 40-45 minutes. Question-answer and discussion methods were used during the training. After the training, the mothers were asked to fill out the same scale again one month later. One month after the training, the mothers were interviewed face-to-face and the scale was filled in again and the changes they made at home were recorded.
  Arms: Educated
Other: Control Group — Mothers in the control group were informed about the research and the 'Informed Consent Form' was signed. The mothers filled out the 'Information Form' and this process took about 15-20 minutes. Mothers were helped when filling out the form and their questions were answered. In addition, mothers were asked to complete the 'Diagnostic Scale of the Mother's Safety Measures for Home Accidents in Children Aged 0-6' by introducing. A month later, they were informed that they had to fill out this scale again. A month later, the mothers were interviewed face-to-face and allowed to fill out the scale again. After the last test, the mothers in the control group were given 'Home Accidents and Prevention Training for Children in the 0-6 Age Group' and the output of the training presentation was distributed.
  Arms: Uneducated

SUMMARY:
The aim of this research is to examine the effect of education for home accidents given to mothers with mentally disabled children in the age group of 0-6.

DETAILED DESCRIPTION:
This study was conducted to examine the effects of education on home accidents given to mothers of mentally disabled children aged 0-6. The sample of the study consisted of 83 mothers of mentally disabled children aged 0-6 registered in four special education centers in Kocaeli province between May 2023 and June 2024 (education group: 40 mothers; control group: 43 mothers). Research data were collected using the Information Form and the Scale for Diagnosing Mothers' Safety Precautions for Home Accidents in 0-6 Year Old Children. The mothers in the education and control groups were informed about the study, their written consent was obtained, and they were asked to fill out information forms. The mothers in the education group were given a single, 45-minute face-to-face education on preventing home accidents. The Mothers' Safety Measures for Home Accidents in Children aged 0-6 were administered the Scale before and one month after the training. The mothers in the control group did not receive any training; the Scale for Identifying Mothers' Safety Precautions for Home Accidents in Children Aged 0-6 was administered during the first interview and again one month later.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with mentally disabled children aged 0-6
* Mothers who agree to participate in the research
* Mothers who agree to be contacted after 1 month for the post-test
* Mothers who know and speak Turkish at the native level

Exclusion Criteria:

* Mothers with mentally disabled children over the age of 6
* Mothers who do not agree to participate in the study
* Mothers who do not agree to be contacted after 1 month for the post-test
* Mothers with mental disabilities
* Mothers who do not know or speak Turkish at the native level

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The Scale for Diagnosing the Safety Measures of the Mother for Household Accidents in Children Aged 0-6 | Before the training and one month after the training.
  The scale developed by Çınar and colleagues evaluates the safety precautions taken by mothers of children aged 0-6 to protect their children from home accidents (burns, falls, poisoning, sharp-edged injuries, foreign object aspiration, drowning, electric shocks). The Scale for Identifying Mothers' Safety Precautions for Home Accidents in Children Aged 0-6 consists of a total of 40 items, with 34 positive and 6 negative statements. Each item is scored between 1-5 on the five-point Likert-type scale. While the items containing positive statements always receive 5 points, often 4 points, sometimes 3 points, rarely 2 points, and never 1 point, the items containing negative statements receive 6, 9, 23, 26, 30, and 40 never 5 points, rarely 4 points, sometimes 3 points, often 2 points, and always 1 point. The minimum score of the scale is 40 and the maximum score is 200. The Croncbach alpha internal consistency coefficient value is 0.82.

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)